CLINICAL TRIAL: NCT02778243
Title: Sexual Steroids: Relationship Between Serum and Prostatic Tissue Level
Acronym: STERPROSER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014/01; 2014-A00706-41 (Other: ANSM)
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2016-11

CONDITIONS: Urinary Bladder Neoplasms; Prostate Hyperplasia
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bladder cancer (Experimental): ▪ Patients justifying prostatectomy together with the bladder (radical cystectomy for bladder cancer).
  Interventions: Biological: steroids concentrations determination
- benign prostate hyperplasia (Other): ▪ Patients with benign prostate hyperplasia who justified a prostatectomy.
  Interventions: Biological: steroids concentrations determination

INTERVENTIONS:
Biological: steroids concentrations determination

SUMMARY:
Patients followed in the Foch Hospital Urology Department (Suresnes): Patients justifying a prostatectomy.

* Patients justifying prostatectomy together with the bladder (radical cystectomy for bladder cancer).
* Patients with benign prostate hyperplasia who justified a prostatectomy. Compare serum sexual steroid concentrations and intra-tissue on healthy prostates and prostate adenoma, assess concentrations intra-tissue sex steroids on cancer metastasis prostate specific blood sample under study (30mL) will be performed preoperatively in Patients followed in Foch Hospital Urology Department (Suresnes), and a Removal of a fragment of prostate tissue or metastasis will be analyze.

Aim is to compare serum concentrations of sexual steroids and intra-tissue on healthy prostates and prostate adenomas compared to concentrations measured in patients operated for prostate cancer.

DETAILED DESCRIPTION:
Steroids concentration will be determined using Gas chromatography-mass spectrometry. The analyzed steroids are :

FSH :Mul/ml LH: mUI/ml SHBG: µg/ml BT: ng/ml TT: ng/ml DHT: ng/ml DHEA: ng/ml D5: ng/ml D4: ng/ml E1: pg/ml E2 : pg/ml DHEA-S : µg/dl

ELIGIBILITY:
Inclusion Criteria:

* Men aged over 18 years
* Surgical indication justifying protatique prostatectomy, or complete prostatocystectomie, or removal of a metastasis of prostate cancer.
* Patients affiliated to a social security scheme or benefiting from such a regime.
* Patients who have given their consent to participate in writing

Exclusion Criteria:

* Patient received local therapy or hormonal treatment (LHRH analogue, therapy blocking androgen receptors) before surgery.
* Treatment reductase inhibitors 5ARI ongoing or stopped for less than 3 months before the intervention.
* Patient included in another clinical trial inconsistent with the conduct of this research.
* Patient receiving treatment that could interfere with hormone levels (Prednisone, Ketoconazole, Abiraterone, Finasteride, Dutasteride).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-11-12 (Actual); Study Completion 2016-11-12 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of sexual steroids and intra-tissue on healthy prostates | 30 minutes
  A bio-informatical analysis will be performed to compare steroids concentrations profiles in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Botto, PhD, Principal Investigator — Urologie Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No